CLINICAL TRIAL: NCT04185961
Title: A Double-blind Pilot Study to Determine the Optimal Negative Pressure of EVERA-RAPHA for Non-invasive Breast Augmentation in Women
Brief Title: Pilot Study to Determine the Optimal Negative Pressure for Non-invasive Breast Augmentation in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GNSD_EVRP_2019
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Breast Hypoplasia

STUDY DESIGN:
Intervention Model Description: EVERA-RAPHA with 60 mmHg: EVERA-RAPHA apply 15 minutes with 60mmHG every day for 4 weeks EVERA-RAPHA with 100 mmHg: EVERA-RAPHA apply 15 minutes with 100mmHG every day for 4 weeks
Who Masked: Participant, Outcomes Assessor
Masking Description: A Double-blind Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVERA-RAPHA with 60mmHG (Experimental): EVERA-RAPHA apply 15 minutes with 60mmHG every day for 4 weeks
  Interventions: Device: EVERA-RAPHA with 60mmHG
- EVERA-RAPHA with 100mmHG (Experimental): EVERA-RAPHA apply 15 minutes with 100mmHG every day for 4 weeks
  Interventions: Device: EVERA-RAPHA with 100mmHG

INTERVENTIONS:
Device: EVERA-RAPHA with 60mmHG — Apply EVERA-RAPHA with 60mmHG for 4weeks
  Arms: EVERA-RAPHA with 60mmHG
Device: EVERA-RAPHA with 100mmHG — Apply EVERA-RAPHA with 100mmHG for 4weeks
  Arms: EVERA-RAPHA with 100mmHG

SUMMARY:
Aim is to investigate optimum pressure and evaluate safety and effectiveness of EVERA-RAPHA for breast augmentation

DETAILED DESCRIPTION:
1. Subjects who voluntarily signed a consent form and met all inclusion / exclusion criteria should enroll in this study.
2. Subjects enrolled in the study will be randomized and assigned to either Group1 or Group2 in a 1: 1 ratio.
3. Apply EVERA RAPHA for 4 weeks

3. Measure breast circumference and breast volume at Baseline and 4weeks later 4. Visit after 4 weeks to evaluate safety and effectiveness

ELIGIBILITY:
Inclusion Criteria:

1. A woman over the age of twenty
2. A woman who wants both breast enlargement
3. A person whose difference between chest circumference and lower chest circumference is less than 10 cm.
4. Subject who sign the consent form of the study and agree to participate in the clinical trial
5. Subject who are willing and able to comply with study protocol

Exclusion Criteria:

1. A woman who has a history of great weight-change
2. A case that Breast cancer or mammary tumour found in basic physical examinations
3. A woman with symptoms or history that suggest she has a fibroblastoma, breast pain, periodic congestion, etc.
4. A woman with severe trauma around the breast.
5. A woman with a scar or skin lesion around the breast.
6. A woman with more than breast ptosis of Grade 3 (the nipple is less than 1-3 cm below the breast)
7. A woman with a history of chronic dermatitis, chronic pressure urticaria, contact dermatitis, etc.
8. A woman who disagrees with contraception
9. A woman who has previously undergone a breast reconstruction or breast augmentation
10. A woman with an uncontrolled active infectious disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
change in the breast volume between before and after 4 weeks in test group 1 and test group 2 respectively. | Baseline and after 4 weeks
  change in the breast volume between before and after 4 weeks of wearing the medical device in test group 1 and test group 2 respectively.

SECONDARY OUTCOMES:
change in the breast circumference between before and after 4 weeks in test group 1 and test group 2 respectively. | Baseline and after 4 weeks
  change in the breast circumference between before and after 4 weeks of wearing the medical device in test group 1 and test group 2 respectively.
difference the mean breast volume between test group 1 and test group 2 | Baseline and after 4 weeks
  difference the mean breast volume between test group 1 and test group 2
difference the mean breast circumference between test group 1 and test group 2 | Baseline and after 4 weeks
  difference the mean breast circumference between test group 1 and test group

CONTACTS AND LOCATIONS:
Overall Officials: Chan Yeong Heo, Doctor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Bundang,Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No